CLINICAL TRIAL: NCT05348746
Title: ERASE - Rise Against Malaria Project - Support for Malaria Prevention, Diagnosis and Treatment in the Context of the Covid-19 Pandemic Among Pregnant Women in Northern Uganda: a Prospective Observational Study
Brief Title: ERASE - Impact of COVID-19 on Malaria Control
Acronym: ERASE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Doctors with Africa - CUAMM (Other)
Collaborators: University of Bari "Aldo Moro", Bari Italy (Unknown); Istituto Superiore di Sanità, Rome, Italy. (Unknown); Catholic University of the Sacred Heart (Other); Doctors with Africa CUAMM, Kampala Uganda (Unknown); Doctors with Africa-Cuamm, Padua, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: Doctors with Africa CUAMM
Record Dates: First submitted 2022-04-10; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Malaria; Malaria in Pregnancy
Keywords: Malaria resistance; COVID 19; Malaria in Pregnancy
MeSH Terms: conditions — Malaria; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Target P. falciparum drug resistance genes: Pfk13 propeller, Pfdhfr and Pfdhps. The polymorphisms analysis of the propeller domain of the Pfk13 gene will be performed by PCR amplifications and subsequent sequencing. Analysis of Pfdhfr gene at codons 51, 59, 108 and Pfdhps gene at codon positions 436, 437, 540, 581, 613 will be done by means of amplifications and subsequent Sanger sequencing. he obtained sequences will be compiled and analyzed by Accelrys DS Gene software. PlasmoDB gene identification no. PF3D7_1343700 (P. falciparum 3D7 strain) will be used as reference in the numbering of nucleotide and amino acid positions. Molecular studies will be performed only for research purposes and will have no impact on the clinical management of study patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Advanced Analysis of Polymorphism — Assessment of Plasmodium falciparum drug resistance. Target P. falciparum drug resistance genes: Pfk13 propeller, Pfdhfr and Pfdhps. The polymorphisms analysis of the propeller domain of the Pfk13 gene will be performed by PCR amplifications and subsequent sequencing. Analysis of Pfdhfr gene at codons 51, 59, 108 and Pfdhps gene at codon positions 436, 437, 540, 581, 613 will be done by means of amplifications and subsequent Sanger sequencing. Molecular studies will be performed only for research purposes and will have no impact on the clinical management of study patients.

SUMMARY:
Objective: Measure incidence of malaria and malaria-related outcomes, evaluating potential impact of the SARS-CoV2 epidemic and of antimalarial resistance in Oyam and Kole district, Uganda with focus on pregnant women.

Study design: Facility-based, prospective, observational study.

Study population: All pregnant women at any gestational age presenting to the Aber Hospitals during the study period both at the emergency department or the Ante-Natal Care (ANC) clinic will be eligible to participate in this study.

Methods: Women will be recruited at ANC visits and at the emergency department and screened against the inclusion criteria. Women will be followed until delivery and evaluated during the consecutives ANC visits. Outcomes will be assessed at the delivery or/and at the discharge if admitted to the hospital for any other causes related with the pregnancy or the malaria. Also, a subpopulation of nonpregnant individuals diagnosed with malaria will be recruited for resistance detection.

Main study parameters/primary endpoints: Incidence of malaria and malaria-related adverse outcomes; impact of the COVID-19 pandemic on malaria care; prevalence of antimalarial resistance against artemisinin derivatives and sulphadoxine-pyrimethamine.

DETAILED DESCRIPTION:
1. INTRODUCTION

1.1. Malaria epidemiology and global trends Globally, there were an estimated 241 million malaria cases in 2020 in 85 malaria endemic countries, increasing from 227 million in 2019, with most of this increase coming from countries in the WHO African Region.

Although it still represents a major threat for public health, over the last twenty years tremendous progress has been made on malaria control, averting an estimate of 1.5 billion cases and saving 7.6 million lives. Malaria mortality fell by 60% over the period from 2000 to 2019, especially in Africa, where political commitment, ignited by the 2000 Abuja declaration has been the key to success. Along with strong political leadership, these data outline the potential benefit in malaria control and prevention brought by public health programs. However, despite the astonishing results achieved in the last two decades, in 2020, COVID-19 pandemic added a crucial challenge in the fight against the disease, posing a major risk for Low and Middle Income Countries (LMICs). In fact, in sub-Saharan countries, along with the substantial danger posed directly to the already fragile healthcare systems, malaria control has been threatened by supply-chain interruptions and by individual decision-making adaptation. Indeed, malaria control relies heavily on individual choice to seek care, and early messaging targeted on reducing SARS-CoV2 transmission advised people to stay home in case of fever. According to geostatistical models, these factors may contribute to an estimated increase, in a worst-case scenario, of 21% malaria cases and nearly double malaria-related deaths in the upcoming years. Furthermore, the true COVID-19 burden in sub-Saharan countries is unknown and, according to seroprevalence studies, it is likely to be largely underestimated . All these factors, according to the latest WHO World Malaria Report, contributed to a reverse of the reducing trend in malaria case incidence (59 cases per 1000 people at risk in 2020, compared to 56 in 2019) and malaria deaths, that passed from 534,000 in 2019 to 602,000 in 2020.

Other substantial challenges towards malaria eradication are drug-resistance, acquisition of mutations impairing diagnosis - especially those affecting the sensitivity of rapid-diagnostic tests - access to treatment and supply of malaria prevention tools such as insecticide-treated mosquito nets (ITN), Indoor Residual Spraying (IRS), Seasonal Malaria Chemoprevention (SMC) and Intermittent Preventive Treatment for pregnant women (IPTp).

1.3 RESEARCH QUESTIONS

1. How COVID-19 pandemic impacted malaria care and malaria-related prevention attitudes among pregnant women in Oyam and Kole districts?
2. What is the prevalence of clinical resistance against SP and artemisinin in Oyam and Kole districts?
3. How COVID-19 pandemic and antimalarial resistance impacted malaria-related outcomes in pregnant women?

1.4 OBJECTIVES 1.4.1 Main Objective The general aim of the study is to assess the impact of Antimalarial Resistance and COVID-19 Pandemic on Malaria Prevention, Diagnosis and Treatment among Pregnant Women in Northern Uganda.

1.4.2 Specific Objectives

1. Assess the impact of the COVID-19 pandemic on malaria prevention and control practices for pregnant women in terms of: i) access to antenatal care visits, ii) administration of IPTp, iii) healthcare seeking behavior in case of fever, iv) healthcare provider compliance with national and international guidelines, v) supply and use of insecticide-treated nets and indoor residual spraying in Oyam and Kole district for the period March 2022 to June 2023.
2. Assess incidence of symptomatic and severe malaria in the study cohort in Oyam and Kole district for the period March 2022 to June 2023.
3. Evaluate the determinants of malaria prevention and control compliance in pregnant women in Oyam and Kole district for the period March 2022 to June 2023.
4. Assess incidence of malaria-related adverse maternal and fetal outcomes (maternal anemia, maternal mortality, abortion, low birthweight, prematurity, perinatal mortality, placental malaria) in Oyam and Kole district for the period March 2022 to June 2023.
5. Assess ideation and knowledge regarding SARS-CoV2 infection and malaria among preganant women in Oyam and Kole district for the period March 2022 to June 2023.
6. Assess the prevalence of asymptomatic P. falciparum infection in the study cohort in Oyam and Kole district for the period March 2022 to June 2023.
7. Evaluate the status of circulating dhfr and dhps haplotypes by describing polymorphisms in the P. falciparum dhfr and dhps genes and estimate the prevalence of dhfr / dhps combined mutant haplotypes associated with pyrimethamine and sulfadoxine resistance in the study cohort and in a population of patients diagnosed with malaria in Oyam and Kole district for the period June 2022 to May 2024.
8. Evaluate the emergence and local spread of artemisinin resistance by means of the analysis of polymorphisms in the P. falciparum kelch 13 gene in the study cohort and in a population of patients diagnosed with malaria in Oyam and Kole district for the period June 2022 to May 2024.

   2.0 METHOD AND MATERIALS 2.1 STUDY DESIGN: This will be a health facility based prospective observational study, using quantitative methods of data collection. Semi-structured questionnaires will be administered to collect the data. The data will be collected prospectively, following a cohort of pregnant women presenting to antenatal care visits until delivery. Also, a subpopulation of nonpregnant individuals diagnosed with malaria will be recruited for resistance detection. Collected data will explore the attitude towards malaria prevention during the COVID-19 pandemic, in terms of access to antenatal care visits, administration of IPTp, healthcare seeking behaviour in case of fever, use of insecticide-treated nets and Indoor residual spraying, ideation and knowledge in regard to SARS-CoV2 infection and malaria.

   2.2 STUDY SETTING The study will be conducted at Aber hospital and selected Health Facilities in Oyam and Kole districts, Lango region. Both the hospital and the district Health Centers are managed by the NGO Doctors with Africa CUAMM.

   St. John's Hospital Aber is a private, non-profit, community hospital owned by the Roman Catholic Diocese of Lira and is accredited by the Uganda Catholic Medical Bureau. The hospital is administered by Sisters of Mary, Mother of the Church, a religious congregation. The hospital has a capacity of 220 beds. Aber Hospital has annual outpatient department attendance of 27,827 contacts, 6,800 admissions with a bed occupancy rate of about 40% and 1,700 average annual maternal deliveries with a cesarean section rate of 21%.

   Oyam district it is located in the Northern part of Uganda. It has it total population of 366,200 people. It is bordered by the Districts of Gulu in the North, Kiryandongo in the South West, Nwoya in the West, Apac in the South and Kole in the East. The district comprises of 12 sub counties i.e. Loro, Minakulu, Aber, Acaba, Ngai, Iceme, Otwal, Abok, Myene, Aleka, Kamdini, and Oyam Town Council. Kole District is bordered by Lira District to the east, Apac District to the south and Oyam District to the west and north. Kole, the district capital, is located approximately 28 kilometres (17 mi), by road, northwest of Lira, the largest city in the sub-region. Kole district is subdivided into the following sub-counties: Aboke, Akalo, Alito, Ayer, Bala, Okwerodot, Ayer Town Council.

   2.3 SAMPLING PROCEDURE AND SAMPLE SIZE ESTIMATION 2.3.1 Sample size estimation Resistance detection

   Considering that:
   * the expected prevalence of parasitaemia among asymptomatic pregnant women is 5%
   * the expected prevalence of parasitaemia among pregnant women who are febrile is 13%
   * in 2019, the prevalence of P. falciparum carrying gene polymorphisms associated with resistance was 20% for artemisinin derivates and 16% for SP.

   In order to estimate the proportion positive for P. falciparum with a 2% absolute precision, at a power of 80% and a 5% level of significance (two sided), a minimum of 800 pregnant women will be required, allowing for a 10% loss to follow-up. The investigators need to recruit 1200 - 1400 women with unknown parasitological status to detect around 20 resistances, even considering an increasing trend.

   To support the achievement of the minimum sample size, the researcher need to recruit a subpopulation of nonpregnant, microscopically confirmed malaria patients from Aber Hospital. This additional recruitment will be performed by consecutive enrollment until the attainment of the minimum sample size of 300 microscopically confirmed, P. falciparum infected samples.

   Cohort of pregnant women Study population will be recruited by consecutive sampling, from 1st May 2022 to 30 June 2023.

   2.3.2 Sampling procedure

   The health facilities will be selected by purposive sampling. The sampling will be based on the following criteria:
   * laboratory capacity
   * presence of an experienced microscopist
   * antenatal care visit volumes of at least 50 visits per month
   * quality of service as per periodic CUAMM assessment

   2.3.3 Selection of participants Participants coming to the sampled healthcare facilities who meet the eligibility criteria will be included in the study. Consecutive enrollment of participants will be undertaken up to when the minimum sample size required for the study will be met.

   2.7 STUDY PROCEDURES AND TIMELINE

   2.7.1 Study procedures Microscopy Thick and thin blood smears will be stained with 2% Giemsa and read by experienced laboratory technologists. Parasite densities will be calculated by counting the number of asexual parasites per 200 leukocytes (or per 500 leukocytes, if the count is <10 asexual parasites/200 leukocytes), assuming a leukocyte count of 8,000/µl. A blood smear will be considered negative when the examination of 100 high power fields does not reveal asexual parasites. Gametocytemia will also be determined from thick smears. Thin smears w1ill be used for parasite species identification.

   Molecular diagnosis and Plasmodium species confirmation The blood samples of the patients will be collected using filter paper (Whatman 3 MM) during admission to the healthcare facility. The dried blood spots (DBSs) will be collected through a finger prick (three drops of blood per participant) on filter papers which will be dried and kept in plastic bags with desiccant and stored in boxes in a cool dry place at room temperature before being transferred at the ISS for molecular diagnosis and drug resistance analysis.

   Shipment of the Blood samples The collected blood samples will be shipped to Italy for advanced Polymorphism analysis. During shipment, all the samples will be stored in a dry, cool place at room temperature to the Italian National Institute of Health (Istituto Superiore di Sanità, ISS).

   Advanced Analysis of Polymorphism Total genomic DNA will be extracted from filter blots (3MM Whatman) using the PureLink Genomic DNA Kits-Invitrogen, according to the manufacturer's recommendation. Parasite identification is based on nested PCR assay targeting the 18S rRNA gene. The 18S rRNA gene is used as a target since it contains both highly conserved and variable regions for each Plasmodium species. The genus-specific PCR will be followed by Plasmodium species-specific PCR amplification. Amplicons from the second PCR will be separated by electrophoresis on a 2% agarose gel and stained with ethidium bromide for visualization using ultraviolet trans-illumination. The presence of parasitaemia will be confirmed when the expected band size corresponding to P. falciparum, P. vivax, P. malariae and or P. ovale will be identified.

   Assessment of Plasmodium falciparum drug resistance. Target P. falciparum drug resistance genes: Pfk13 propeller, Pfdhfr and Pfdhps. The polymorphisms analysis of the propeller domain of the Pfk13 gene will be performed by PCR amplifications and subsequent sequencing. Analysis of Pfdhfr gene at codons 51, 59, 108 and Pfdhps gene at codon positions 436, 437, 540, 581, 613 will be done by means of amplifications and subsequent Sanger sequencing. Commercial oligonucleotide primer pairs for Pfk13 will be obtained based on the published article by Taylor et al., whereas for the analysis of dhfr and dhps genes primer pairs will be obtained based on the published article by Menegon et al. [31]. The obtained sequences will be compiled and analyzed by Accelrys DS Gene software. PlasmoDB gene identification no. PF3D7_1343700 (P. falciparum 3D7 strain) will be used as reference in the numbering of nucleotide and amino acid positions. Molecular studies will be performed only for research purposes and will have no impact on the clinical management of study patients.

   To enhance local capacity building, one laboratory person from Aber hospital will attend a two weeks exposure at the reference laboratory in Italy.

   Study time points TIME POINT STUDY PROCEDURES AND DATA COLLECTION RECRUITMENT (ANC VISIT) - Full questionnaire administered by a trained health care worker to collect information on demographic (eg. age, area of residence), socioeconomic factors (eg. education, occupation), number and outcome of previous pregnancies, date of last menstruation, bed net ownership and use, adherence to malaria chemoprevention, reasons for non-adherence, malaria behaviors, barriers to administration of IPTp, use of ITNs, perceived impact of COVID-19 will be administered.
   * Clinical examination assessing the general wellbeing and nutritional status of the woman, along with routine measurements (including weight, height, auscultation, blood pressure and temperature). Gestational age will be assessed, when available, by obstretic ultrasound and, if unavailable, by pelvis examination performed by experienced midwives
   * Collection of blood sample that will be analyzed as follows:

     * Malaria diagnostic test with microscopy and, when positive, parasite count. Positive samples will be sent to the ISS. Molecular diagnosis will be performed to confirm microscopy results and to discriminate between Plasmodium species. Plasmodium falciparum positive samples will be analyzed for detection of single nucleotide polymorphisms in P. falciparum genes associated with artemisinin and SP resistance. Women diagnosed with malaria will be treated and followed according to Uganda Clinical Guidelines, and parasitemia will be reassessed at day 3.
     * HIV diagnostic test.
     * Hemoglobin levels. All women found to be HIV+ at study entry will be referred for further evaluation and treatment.

   ANC VISITS
   * Physical examination
   * Follow-up survey, investigating history of fever, malaria-related prevention attitudes (compliance with IPTp, use of ITN) and eventual barriers in care-seeking due to the COVID-19 pandemic.
   * Malaria diagnostic test with microscopy and, when positive, parasite count. Positive samples will be sent to the ISS. Molecular diagnosis will be performed to confirm microscopy results and to discriminate between Plasmodium species. Plasmodium falciparum Positive samples will be analyzed for detection of single nucleotide polymorphisms in P. falciparum genes associated with artemisinin and SP resistance. Women diagnosed with malaria will be treated and followed according to Uganda Clinical Guidelines, and parasitemia will be reassessed at day 3.

   ANY SPONTANEOUS VISITS TO THE HOSPITAL RELATED WITH PREGNANCY AND/OR MALARIA
   * standardized history
   * physical exam including temperature, pulse, and blood pressure measurement.
   * Participants who are febrile (tympanic temperature > 38.0˚C) or report history of fever in the past 24 hours will have blood obtained by finger prick for a thick blood smear. If the thick blood smear is positive, the patient will be diagnosed with malaria. If the thick blood smear is negative, the patient will be managed by study physicians for a non-malarial febrile illness. If the patient is afebrile and does not report a recent fever, a thick blood smear will not be obtained, except when following routine testing schedules.
   * In patients with positive microscopy for P. falciparum, the first, pre-therapy blood sample collected as DBS will be sent for molecular diagnosis confirmation and for genetic analysis of antimalarial resistance to ISS. Furthermore, in those patients, parasitemia will be reassessed at day 3, as per WHO protocol.
   * Recruitment of the subpopulation of non-pregnant individuals will be undertaken at this time point.

   DELIVERY
   * Delivery information: study staff will document details of the delivery, including date and time, type of delivery, estimated blood loss and any maternal, obstetrical or neonatal complications.
   * Fetal outcome.
   * Infant information: Apgar score and birth weight with calibrated scales. At the time of delivery, women will undergo repeat rapid HIV testing based on national guidelines. If women are found to have become HIV-infected during pregnancy, both the mother and their newborn will be withdrawn from the study and immediately referred for care following local prevention of mother-to-child transmission guidelines.

   2.8 DATA COLLECTION AND MANAGEMENT 2.8.1 Data collection tools Data will be collected using semi-structured questioners and managed using REDCap electronic data capture tools hosted at "Catholic University of the Sacred Heart", Rome, Italy, REDCap (Research Electronic Data Capture) is a secure, web-based software platform designed to support data capture for research studies, providing 1) an intuitive interface for validated data capture; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for data integration and interoperability with external sources.

   2.8.2 Management of the Anti-malarial resistance data Data will be recorded on standard study data collection forms and will be reviewed for accuracy and completion. Upon resolution of data forms errors/missing values, the form will be ready for data entry. The obtained results will be entered into a database. A database will be developed to accommodate data entry and management of the study's data. The database will be created with a standard data management software package, such as Microsoft Access. A file for each study form will be created. The analysis of the sequenced samples will produce a number of standardized reports: separate Excel datasheets and maps for associated drug resistance SNPs and all other SNPs (exonic and intronic). In addition, individual sample variant call format (VCF) files will be generated.

   2.8.3 COVID-19 Mitigation Measures:

   The investigators know that the COVID-19 risk will continue for most of the study duration. All study procedures including data collection and management activities will be implemented with this understanding in mind and the following COVID-19 risk mitigation measures will be followed:
   * All study staff will be oriented on COVID-19- standard operation procedures (SOPs) as communicated by Ministry of Health (MOH)
   * The orientation meetings will follow the MOH recommended number of participant in line with the COVID-19 prevention protocols.
   * The investigators shall regularly use the zoom platform for online meetings to update on study progress across the study sites
   * The study staff and participants will be provided with COVID-19 personal protective equipment (Mask, Hand sanitisers, and hand washing soap) to use when implementing the study activities
   * COVID-19 prevention protocols will be published, displayed and followed in all study activity areas and attention of participants will be drawn to these protocols as part of the introductory communication also to ensure continuation of access to essential services.
   * All study staff and participants will be provided with adequate information and encouraged to take the COVID-19 vaccination as recommended by MOH

   2.11 ETHICAL CONSIDERATIONS A study protocol will be submitted for approval to the Lacor Hospital research Ethics committee and the Uganda National Council of Science and Technology (UNCST). Pregnant women will be asked for written informed consent to participation to the study. We shall administer consent at two levels; first we shall administer and obtain consent for participation in the study and thereafter consent for collection and transportation of blood samples to Italy. The blood samples collected will be used only for the purpose of this study and will not be stored beyond the current study project. All unprocessed blood samples will be destroyed from the department of infectious disease, university of Bari-Italy as biological sanitary waste, at the end of the project. The same standard of care will be guaranteed to all pregnant women irrespectively of participation. The dignity of study participants will be guaranteed by the investigators, as well data confidentiality and the right to withdraw data and/or biological samples at any time. Consent to pregnant women and to mature and emancipated minors will be obtained according to Uganda Human Subjects Protection Guidelines.

   For all malaria positive samples processed for molecular analysis in the present study, identifying information will be removed to provide appropriate protection of medical confidentiality and privacy. In this way, sensitive data cannot be linked or re-linked with identifiable human subjects, making anonymous each sample processed.

   The polymorphisms analysis of the propeller domain of the Pfk13 gene will be performed by advanced amplifications techniques and subsequent Sanger sequencing in a highly specialized scientific laboratory. The blood samples collected in this study will be sent to a laboratory in the University of Bari, Italy, in order to have access to the latest Pfk13 gene amplification techniques. To enhance local capacity building one laboratory staff from Aber hospital will be supported to attend a two weeks exposure at the reference laboratory in Italy Clearance for blood sample shipment to Italy: Approval for sample transportation will be obtained from UNCST before shipment of any blood samples to Italy. A request for transfer of the blood samples will be made in writing to the executive secretary of UNCST. This will be accompanied by a material transfer agreement (MTA) between Pope John hospital Aber (the transferor), Doctors with Africa CUAMM (the study partner), and the Department of Infectious Diseases-University of Bari (the recipient) . The exact specification of the transfer conditions and the approved study protocol will as well be submitted to UNCST with the request for the transfer of the blood samples.

ELIGIBILITY:
Inclusion Criteria: All pregnant women at any gestational age presenting to the Aber Hospitals during the study period both at the emergency department or the Ante-Natal Care (ANC) clinic will be eligible to participate in this study.

Inclusion criteria will be:

•. Pregnancy confirmed by positive urine pregnancy test or intrauterine pregnancy by ultrasound;

* Provision of informed consent;
* Agreement to come to the study clinic for any febrile episode or other illness;
* Plan to deliver in the hospital

Exclusion Criteria:

• Ongoing labor or delivery

Non-pregnant subpopulation

Inclusion criteria for this population will be:

* microscopically confirmed diagnose of malaria ;
* provision of informed consent;
* agreement to avoid antimalarial medications given outside the study protocol;
* agreement to be re-assessed for parasitemia at day 3 Exclusion Criteria
* too ill to participate in the study according to clinician judgment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Target population All pregnant women living in Oyam and Kole districts. Accessible population Pregnant women in Oyam and Kole district coming for antenatal care in Aber Hospital and selected Healthcare facilities during the study period March 2022 to June 2023.
  Non-pregnant subpopulation For epidemiological assessment of resistance against sulfadoxine-pyrimetamine and artemisinin derivatives, a sub-population of individuals diagnosed with microscopically confirmed malaria in Aber hospital will be also recruited. This population is necessary to reach an adequate sample size for resistance detection.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Impact of COVID 19 in Malaria care | 12 months
  The investigators using retrospective data from 2018-2019 (pre COVID era) to 2020-2021 (COVID era) will evaluate i) access to antenatal care visits, in Oyam and Kole district for the period March 2022 to June 2023.
  Antenatal care visits: The percentage of women aged 15-49 with a live birth in a given time period that received antenatal care four or more times. Due to data limitations, it is not possible to determine the type of provider for each visit. Numerator: The number of women aged 15-49 with a live birth in a given time period that received antenatal care four or more times. Denominator: Total number of women aged 15-49 with a live birth in the same period.
Impact of COVID 19 in Malaria care | 12 months
  The investigators using retrospective data from 2018-2019 (pre COVID era) to 2020-2021 (COVID era) will evaluate ii) IPTp (intermittent preventive treatment) coverage in Oyam and Kole district for the period March 2022 to June 2023.
  IPTp (intermittent preventive treatment) coverage will be study and define in two ways:
  * the proportion of women who had received at least one ITP dose during their pregnancy, designated as "ITP coverage-at least one dose";
  * the proportion who had received both ITP doses recommended, designated as "ITP coverage-two doses."
Incidence of symptomatic and severe malaria in the study cohort | 12 months
  Assess incidence of symptomatic and severe malaria in the study cohort in Oyam and Kole admitted to Aber Hospital and health district for the period March 2022 to June 2023.
Determinants of malaria prevention | 12 months
  Due to survey KAP (knowledge, attitude and practice) for pregnant women admitted in antenatal clinic , the investigators will evaluate the determinants of malaria prevention and control compliance in pregnant women in Oyam and Kole district for the period March 2022 to June 2023

SECONDARY OUTCOMES:
Prevalence of Plasmodium species resistant | 12 months
  The investigators will evaluate the prevalence of resistance against SP derivatives in a population of malaria cases diagnosed in the study centers during the study period.
  Parasite identification is based on nested PCR assay targeting the 18S rRNA gene. The 18S rRNA gene is used as a target since it contains both highly conserved and variable regions for each Plasmodium species. The genus-specific PCR will be followed by Plasmodium species-specific PCR amplification. Amplicons from the second PCR will be separated by electrophoresis on a 2% agarose gel and stained with ethidium bromide for visualization using ultraviolet trans-illumination. The presence of parasitaemia will be confirmed when the expected band size corresponding to P. falciparum, P. vivax, P. malariae and or P. ovale will be identified.
Incidence of maternal and fetal outcome | 15 months
  The researcher will evaluete in pregnant women with Malaria enrolled in the study the incidence of malaria-related adverse maternal and fetal outcomes (maternal anemia, maternal mortality, abortion, low birthweight, prematurity, perinatal mortality, placental malaria) in Oyam and Kole district for the period March 2022 to June 2023
Local spread of P. falciparum polymorphisms | 24 months
  The investigators will evaluate the emergence and local spread of artemisinin resistance by means of the analysis of polymorphisms in the P. falciparum kelch 13 gene in the study cohort and in a population of patients diagnosed with malaria in Oyam and Kole district for the period June 2022 to May 2024.
  The polymorphisms analysis of the propeller domain of the Pfk13 gene will be performed by PCR amplifications and subsequent sequencing. Analysis of Pfdhfr gene at codons 51, 59, 108 and Pfdhps gene at codon positions 436, 437, 540, 581, 613 will be done by means of amplifications and subsequent Sanger sequencing. The obtained sequences will be compiled and analyzed by Accelrys DS Gene software. PlasmoDB gene identification no. PF3D7_1343700 (P. falciparum 3D7 strain) will be used as reference in the numbering of nucleotide and amino acid positions.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Segala FV, Ictho J, L'Episcopia M, Onapa E, De Vita E, Novara R, Olung N, Totaro V, Olal L, Patti G, Bingom C, Farina U, Papagni R, Agaro C, Bavaro DF, Amone J, Dall'Oglio G, Ngole B, Marotta C, Okori S, Zarcone M, Ogwang J, Severini C, Lochoro P, Putoto G, Saracino A, Di Gennaro F. Impact of the COVID-19 pandemic on malaria in pregnancy indicators in Northern Uganda: a joinpoint regression analysis. Pathog Glob Health. 2024 May;118(3):253-261. doi: 10.1080/20477724.2023.2273023. Epub 2023 Oct 23. PMID 37872763
- [Derived] Segala FV, Di Gennaro F, Ictho J, L'Episcopia M, Onapa E, Marotta C, De Vita E, Amone J, Iacobelli V, Ogwang J, Dall'Oglio G, Ngole B, Murri R, Olal L, Fantoni M, Okori S, Putoto G, Severini C, Lochoro P, Saracino A. Impact of antimalarial resistance and COVID-19 pandemic on malaria care among pregnant women in Northern Uganda (ERASE): protocol of a prospective observational study. BMC Infect Dis. 2022 Aug 4;22(1):668. doi: 10.1186/s12879-022-07645-3. PMID 35927713